CLINICAL TRIAL: NCT02280057
Title: Randomized, Cross-over Trial With Metformin in Women With Polycystic Ovary Syndrome
Brief Title: Trial With Metformin in Women With Polycystic Ovary Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Herning Hospital (Other)
Collaborators: GEA A/S Denmark (Unknown)
Responsible Party: Principal Investigator, Finn Friis Lauszus, Senior Consultant, Herning Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2166-00
Record Dates: First submitted 2014-10-28; First posted 2014-10-31 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS; metformin; obesity; randomized controlled trial
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Active Comparator): Metformin 850 mg x 2 in six months
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Placebo 2 tablets daily for six months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Metformin 1500 mg (=2 pills) per day in six months
  Arms: Metformin
Drug: Placebo — 2 pills per day in six months; pills look like metformin pills
  Arms: Placebo

SUMMARY:
The investigators wanted to elucidate the effects of metformin in Polycystic Ovary Syndrome (PCOS) by performing a randomized, double-blinded, placebo-controlled cross-over study.

DETAILED DESCRIPTION:
Eligible women who gave written informed consent were assigned to 6 months of treatment with either 850 mg of metformin or placebo twice daily, followed by a wash-out period of 3 months before cross-over to the alternate treatment for another 6 months. Randomization defining treatment sequence was done at inclusion by random number tables. The appearance of the tablets was identical, and patients and investigators were blinded to treatment allocation. The randomization code was stored in a closed envelope until all participants had finished the treatment. Participants were seen by one of the investigators before inclusion and every second month during treatment periods, always in the morning after an overnight fast of at least 8 h. They were weighed wearing light clothing. Waist circumference was measured at the umbilical level and hip circumference at the trochanter region. Systolic and diastolic blood pressure was measured with a semiautomatic blood pressure monitor and a blood sample was drawn for immediate analysis without respect to bleeding periods. All participants registered their bleeding periods in a calendar during both study periods and the 3 months wash-out period. Calculation of sample size was based on the assumption that at least 50% of the women would experience at least 30% more menstrual periods on metformin than on placebo. Based on a power of 90 (b = 0.10) to detect a significant difference [two-sided P-value of 0.05], the minimum sampling size was calculated to 44 subjects.

We also assumed a 10% drop-out rate, and thus aimed at including 50 women. As drop-out rate quickly rose higher than expected, we decided to include 60 women. In the intention-to-treat analysis, the values of each participant after 6 months of metformin or placebo were compared with the baseline values. Linear regression analysis with the changes in testosterone and homeostasis model assessment (HOMA) index as dependent variables was performed to examine potential relations between the changes. The per protocol analysis included data from participants completing both study periods, i.e. the difference between the values of each participant after placebo and metformin, respectively, was calculated, and a significance test performed on the differences.

ELIGIBILITY:
Inclusion Criteria:

* testosterone value above the upper normal limit and
* oligo- or amenorrhea,

Exclusion Criteria:

* periclimacteric gonadotrophin values,
* hyperprolactinaemia,
* diabetes mellitus,
* impaired thyroid,
* renal or hepatic function,
* hormonal treatment,
* pregnancy,
* lactation or a wish for fertility treatment.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2001-09; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Testosterone (Levels of free testosterone) | six months
  Levels of free testosterone

SECONDARY OUTCOMES:
Insulin sensitivity (measured homeostasis model assessment (HOMA) index) | Six months
  Insulin sensitivity measured homeostasis model assessment (HOMA) index

OTHER OUTCOMES:
Body weight change | Six months
  Body weight changes

CONTACTS AND LOCATIONS:
Overall Officials: Finn F Lauszus, MD, PhD, Principal Investigator — Gyn Dept. Herning Hospital, Herning, Denmark
Locations (1):
- Gynecology Dept. Herning Hospital, Herning, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Trolle B, Flyvbjerg A, Kesmodel U, Lauszus FF. Efficacy of metformin in obese and non-obese women with polycystic ovary syndrome: a randomized, double-blinded, placebo-controlled cross-over trial. Hum Reprod. 2007 Nov;22(11):2967-73. doi: 10.1093/humrep/dem271. Epub 2007 Aug 31. PMID 17766923
- [Result] Trolle B, Lauszus FF, Frystyk J, Flyvbjerg A. Adiponectin levels in women with polycystic ovary syndrome: impact of metformin treatment in a randomized controlled study. Fertil Steril. 2010 Nov;94(6):2234-8. doi: 10.1016/j.fertnstert.2010.01.057. Epub 2010 Mar 2. PMID 20189560
- [Result] Greibe E, Trolle B, Bor MV, Lauszus FF, Nexo E. Metformin lowers serum cobalamin without changing other markers of cobalamin status: a study on women with polycystic ovary syndrome. Nutrients. 2013 Jul 5;5(7):2475-82. doi: 10.3390/nu5072475. PMID 23857221
- [Result] Madsen HN, Lauszus FF, Trolle B, Ingerslev HJ, Torring N. Impact of metformin on anti-Mullerian hormone in women with polycystic ovary syndrome: a secondary analysis of a randomized controlled trial. Acta Obstet Gynecol Scand. 2015 May;94(5):547-51. doi: 10.1111/aogs.12605. Epub 2015 Mar 4. PMID 25736975